CLINICAL TRIAL: NCT02759588
Title: Phase 1b & 2 Study With GL-ONC1 Oncolytic Immunotherapy in Patients With Recurrent or Refractory Ovarian Cancer (VIRO-15)
Brief Title: GL-ONC1 Oncolytic Immunotherapy in Patients With Recurrent or Refractory Ovarian Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genelux Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GL-ONC1-015
Record Dates: First submitted 2016-04-25; First posted 2016-05-03 (Estimated); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Ovarian Cancer; Peritoneal Carcinomatosis; Fallopian Tube Cancer
Keywords: GL-ONC1; oncolytic virus; virotherapy; Viral therapy; immunotherapy; immune therapy; vaccinia; vaccinia virus; Genelux; ovarian cancer; platinum resistant; platinum refractory; peritoneal carcinomatosis; fallopian cancer; cancer; abdominal cancer; imaging; carcinoma; DNA virus; neoplasms; neoplasms by histological type; neoplasms, Glandular and Epithelial; Poxviridae infections; Virus diseases; recurrent ovarian cancer; intermediate platinum-sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Vaccinia; Neoplasms; Carcinoma; Neoplasms by Histologic Type; Neoplasms, Glandular and Epithelial; Poxviridae Infections; Virus Diseases | interventions — Drug Therapy; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GL-ONC1 (Experimental)
  Interventions: Biological: GL-ONC1 alone, or in combination with chemotherapy with or without bevacizumab

INTERVENTIONS:
Biological: GL-ONC1 alone, or in combination with chemotherapy with or without bevacizumab — GL-ONC1 is a genetically-engineered oncolytic vaccinia virus, which is administered via intraperitoneal infusion as multiple doses.

SUMMARY:
The purpose of this study is to determine if GL-ONC1 oncolytic immunotherapy is well tolerated with anti-tumor activity in patients diagnosed with recurrent or refractory ovarian cancer and peritoneal carcinomatosis.

DETAILED DESCRIPTION:
Ovarian cancer (OC) remains the most lethal gynecologic malignancy owing to late detection, intrinsic and acquired chemo-resistance and remarkable heterogeneity. There is an unmet medical need to develop new therapy modalities. In preclinical studies, GL-ONC1, has shown the ability to preferentially locate, colonize and destroy tumor cells in more than 30 different human tumors, including ovarian cancer. GL-ONC1 has been investigated in early stage clinical trials in the United States and Europe via systemic delivery as monotherapy and in combination with other therapies, and via regional delivery as monotherapy. GL-ONC1 treatment was well tolerated across different malignancies, routes of administration, and monotherapy as well as combination therapy protocols. The ability of GL-ONC1 to infect tumor tissue and kill tumor cells was demonstrated. In addition, virus-induced immune activation and favorable anti-tumor immune response have been observed. Evidences of anti-tumor efficacy and clinical benefits have also been documented.

ELIGIBILITY:
Inclusion Criteria:

* Signed, written informed consent.
* High-grade serous (including Malignant Mixed Mullerian Tumor (MMMT) with metastasis that contains high grade epithelial carcinoma), endometrioid, or clear-cell ovarian cancer which includes: (1) platinum-resistant (recurrence or progression in < 6 months) or (2) platinum-refractory (progression while on platinum-based therapy); patient must have failed either at least 2 consecutive therapies or are not eligible for additional cytotoxic therapies (exception is Phase 2 receiving chemotherapy with/without bevacizumab).
* Intermediate platinum-sensitive patients (recurrence of disease 6 to 12 months from last platinum compound treatment): Recurrent ovarian carcinoma with at least four prior individual treatment regimens including at least two separate platinum-based therapies with recurrence from the last platinum-based regimen less than 12 months, who are unwilling or unable to undergo additional platinum-based cytotoxic therapy (this sub-population is not applicable for Phase 2 receiving chemotherapy with/without bevacizumab).
* Performance status ECOG is at 0 or 1, and life expectancy of 6 months
* Has either measurable disease in the peritoneal cavity as defined by RECIST 1.1 (Phase 1b & 2) or has non-measurable disease in the peritoneal cavity (Phase 1b) and can be confirmed by laparoscopy and/or elevated CA-125. Patients who have non-measurable disease that is not identifiable by PET/PET-CT scan, but who have elevated CA-125, and/or ascites, with visible disease confirmed by laparoscopy are also eligible.
* Able to undergo IP injection.
* Adequate renal, hepatic, bone marrow and immune functions.
* Baseline tumor biopsy is required.
* Documented progressive disease status at baseline (Phase 2).

Exclusion Criteria:

* Tumors of mucinous subtypes, or non-epithelial ovarian cancers (e.g., Brenner tumors, Sex-cord tumors).
* Unresolved bowel obstruction.
* Known central nervous system (CNS) metastasis.
* Known seropositivity for HIV or active hepatitis infection.
* History of thromboembolic event within the last 3 months.
* Pregnant or breast-feeding women.
* Smallpox vaccination within 1 year of study treatment.
* Clinically significant cardiac disease.
* Received prior gene therapy or therapy with cytolytic virus of any type.
* Receiving concurrent antiviral agent active against vaccinia virus.
* Have known allergy to ovalbumin or other egg products.
* Have clinically significant dermatological disorders (e.g., eczema, psoriasis, or unhealed skin wounds or ulcers) as assessed by the Investigator.
* Symptomatic malignant ascites and non-manageable pleural effusion.
* Known hypersensitivity to bevacizumab, uncontrolled hypertension, history of stroke, or clinical findings suggestive of excessive risk for GL perforation (uncontrolled peptic ulcer disease, partial small bowel obstruction, etc.) that would make risks of bevacizumab unacceptable in the opinion of the investigator.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05; Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events [Safety and Tolerability] (Phase 1b) | Change from baseline during Treatment and for 30 days following last dose.
  Determine safety and tolerability of administering multiple doses of GL-ONC1 via intraperitoneal catheter by the evaluation of the number of participants with treatment-emergent adverse events (type, frequency, and severity) as assessed by CTCAE 4.03.
Determine Progression-free Survival following Treatment (Phase 2) | From date of registration until the date of first documented disease progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  To assess progression-free survival (PFS) from time of registration until disease
Tumor Marker Cancer Antigen-125 (CA-125) (Phase 2) | Assessed pre-treatment, during treatment at 2- to 3-week intervals and post-treatment assessed up to 24 months.
  To assess anti-tumor response.
Overall Response Rate (ORR) by RECIST 1.1 (Phase 2) | Assessed pre-treatment, during treatment at 6- to 12-week intervals and post-treatment assessed up to 24 months.
  To assess anti-tumor response.

SECONDARY OUTCOMES:
Evaluation of Tumor Response to Treatment (Phase 1b) | Assessed post-treatment at 6 to 12 week intervals or until disease progression or death from any cause, whichever comes first, assessed up to 24 months.
  Evaluate participant's best overall response to treatment with therapeutic intent assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. (i.e., complete response, partial response, stable disease, or progressive disease).
Evaluation of Immune-related Tumor Response | Assessed post-treatment at 6 to 12 week intervals or until disease progression or death from any cause, whichever comes first, assessed up to 24 months.
  Evaluate participants' best overall response to treatment with oncolytic immunotherapy assessed by Immune-related Response Criteria (immune-related complete response, immune-related partial response, immune-related stable disease, or immune-related progressive disease).
CA-125 Response (Phase 1b) | Assessed pre-treatment, during treatment and post-treatment at 6 to 12 week intervals, assessed up to 24 months.
  CA-125 according to the Gynecologic Cancer Intergroup (GCIG) is measured by at least a 50% reduction in CA-125 levels from pre-treatment sample which is confirmed and maintained for at least 28 days. Pre-treatment CA-125 sample must be at least twice the upper limit of normal and obtained within 2 weeks prior to starting treatment.
Determine Progression-free Survival following Treatment (Phase 1b) | From date of registration until the date of first documented disease progression or date of death from any cause, whichever comes first, assessed up to 24 months.
  To assess progression-free survival (PFS) in participant population.
Overall Survival | By medical chart review until death or 3 years from the date of last treatment which ever comes first.
  To determine overall survival (OS) in the participant population.
Clinical Benefit Rate | Approximately 24 months
  Defined as the percentage of patients who have achieved CR + PR + SD greater than or equal to 15 weeks.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Gynecologic Oncology Associates, Newport Beach, California
  - AdventHealth Cancer Institute, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holloway RW, Mendivil AA, Kendrick JE, Abaid LN, Brown JV, LeBlanc J, McKenzie ND, Mori KM, Ahmad S. Clinical Activity of Olvimulogene Nanivacirepvec-Primed Immunochemotherapy in Heavily Pretreated Patients With Platinum-Resistant or Platinum-Refractory Ovarian Cancer: The Nonrandomized Phase 2 VIRO-15 Clinical Trial. JAMA Oncol. 2023 Jul 1;9(7):903-908. doi: 10.1001/jamaoncol.2023.1007. PMID 37227734
- See also: Sponsor's company website — http://www.genelux.com